CLINICAL TRIAL: NCT06156085
Title: Fourteen-Day Vonoprazan-Based Dual Therapy With Amoxicillin as First-Line Helicobacter Pylori Treatment in Comparison With Extended Sequential Therapy: A Randomized Controlled Trial in Taiwan
Brief Title: Fourteen-Day Vonoprazan-Based Dual Therapy With Amoxicillin as First-Line Helicobacter Pylori Treatment in Comparison With Extended Sequential Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fu Jen Catholic University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FJUH112288
Record Dates: First submitted 2023-11-12; First posted 2023-12-05 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2023-11

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Lansoprazole; Clarithromycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VA14 (Experimental): Vonoprazan-Amoxicillin Dual Therapy for 14days
  Interventions: Drug: Vonoprazan and Amoxicillin
- S14 (Active Comparator): Sequential therapy for 14 days
  Interventions: Drug: Lansoprazole, Amoxicillin, Clarithromycin and Metronidazole

INTERVENTIONS:
Drug: Vonoprazan and Amoxicillin — vonoprazan 20 mg and amoxicillin 1000 mg b.i.d. PC for 14days
  Arms: VA14
Drug: Lansoprazole, Amoxicillin, Clarithromycin and Metronidazole — lansoprazole 30 mg + amoxicillin 1000 mg b.i.d. AC for 7 days, followed by the same PPI + clarithromycin 500 mg + metronidazole 500 mg b.i.d. AC for 7 days
  Arms: S14

SUMMARY:
Background：Helicobacter pylori infection is a well-established risk factor for peptic ulcer disease and gastric cancer. It's now a consensus of experts that H.pylori infection should be treated once it is recognized. Extended proton pump inhibitor (PPI)-based sequential therapy as one of the most commonly used first-line regimens provides a satisfactory eradication rate of 90.7% (95% CI, 87.4% - 94.0%). Nevertheless, its complexity of the "sequential" usage is sometimes confusing to the patients and may lead to treatment failure. The emerging new regimen - vonoprazan-based dual therapy, on the other hand, is another appealing choice with simplicity, and low pill burden. However, there's still no evidence regarding the use of vonoprazan-based dual therapy with high-dose amoxicillin (1000mg twice daily) as the first-line regimen in Taiwan. This study aimed to compare the efficacy of the current standard first-line regimen, sequential therapy, with that of vonoprazan-based dual therapy with high-dose Amoxicillin.

Objectives: To compare the efficacy of the current standard first-line regimen, sequential therapy, with that of vonoprazan-based dual therapy, through a randomized controlled trial.

Methods: Patients with H.pylori infection who was over 20 years old and agree to participate in the trial will be recruited. Those who had received H.pylori eradication before, are known to be allergic to any drug used in this trial, are pregnant, or refuse to participate in the trial for any reason will be excluded. We then allocate these patients into two groups randomly - one group receiving vonoprazan-based dual therapy with high-dose amoxicillin (vonoprazan 20 mg + amoxicillin 1000 mg twice daily for fourteen days) and the other receiving extended sequential therapy (lansoprazole 30mg plus amoxicillin 1000mg twice daily for 7 days, followed by lansoprazole 30mg, clarithromycin 500mg, and metronidzole 500mg twice daily for an additional 7 days). Eradication success was evaluated by 13C-urea breath test at least 4 weeks after treatment.

Outcome analysis: The study will be designed as a non-inferiority trial. We anticipate that the two regimens will have comparable efficacy. Besides, we'll also design a questionnaire to evaluate the adverse effects, whether they took the drugs in the right way, and patient's satisfaction of the drug regimen. The vonoprazan dual therapy with high-dose amoxicillin will be anticipated to have fewer adverse effects, better compliance, and better satisfaction.

DETAILED DESCRIPTION:
Background：Helicobacter pylori infection is a well-established risk factor for peptic ulcer disease and gastric cancer. It's now a consensus of experts that H.pylori infection should be treated once it is recognized. Extended proton pump inhibitor (PPI)-based sequential therapy as one of the most commonly used first-line regimens provides a satisfactory eradication rate of 90.7% (95% CI, 87.4% - 94.0%). Nevertheless, its complexity of the "sequential" usage is sometimes confusing to the patients and may lead to treatment failure. The emerging new regimen - vonoprazan-based dual therapy, on the other hand, is another appealing choice with simplicity, and low pill burden. However, there's still no evidence regarding the use of vonoprazan-based dual therapy with high-dose amoxicillin (1000mg twice daily) as the first-line regimen in Taiwan. This study aimed to compare the efficacy of the current standard first-line regimen, sequential therapy, with that of vonoprazan-based dual therapy with high-dose Amoxicillin.

Objectives: To compare the efficacy of the current standard first-line regimen, sequential therapy, with that of vonoprazan-based dual therapy, through a randomized controlled trial.

Methods: Patients with H.pylori infection who was over 20 years old and agree to participate in the trial will be recruited. Those who had received H.pylori eradication before, are known to be allergic to any drug used in this trial, are pregnant, or refuse to participate in the trial for any reason will be excluded. We then allocate these patients into two groups randomly - one group receiving vonoprazan-based dual therapy with high-dose amoxicillin (vonoprazan 20 mg + amoxicillin 1000 mg twice daily for fourteen days) and the other receiving extended sequential therapy (lansoprazole 30mg plus amoxicillin 1000mg twice daily for 7 days, followed by lansoprazole 30mg, clarithromycin 500mg, and metronidzole 500mg twice daily for an additional 7 days). Eradication success was evaluated by 13C-urea breath test at least 4 weeks after treatment.

Outcome analysis: The study will be designed as a non-inferiority trial. We anticipate that the two regimens will have comparable efficacy. Besides, we'll also design a questionnaire to evaluate the adverse effects, whether they took the drugs in the right way, and patient's satisfaction of the drug regimen. The vonoprazan dual therapy with high-dose amoxicillin will be anticipated to have fewer adverse effects, better compliance, and better satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with naive H. pylori infection
2. Subjects with over 20 years old

Exclusion Criteria:

1. Younger than 20 years old
2. Ever received H. eradication therapy
3. ever received total or subtotal gastrectomy in the past
4. Severe chronic disease, such as end stage renal disease, liver cirrhosis, incurable malignant tumors
5. Women who are pregnant or breastfeeding
6. Those who are not suitable to receive study drugs: such as a history of allergies to study drugs or serious side effects, etc.
7. Patient with estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 mt2

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
primary outcome is the eradication rate in the first-line treatment | Up to 8-12 weeks
  At least 6 weeks after the end of treatment, the carbon 13-breath test will be used to evaluate whether the eradication is successful. The eradication rate in each group will be presented as "%

SECONDARY OUTCOMES:
The secondary outcomes are the compliance, frequency of adverse events | Up to 8-12 weeks
  After eradication treatment, participants will go back to the outpatients clinics to evaluate whether they take all of or > 80% drugs. The investigators will also record any side effect associated with treatment, such as skin rash, dizziness, headache, taste distortion, and etc. The severity grading include "none", "mild", "moderate"

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yang Chang, PhD, Study Chair — Fu Jen Catholic University Hospital, Taiwan
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No